CLINICAL TRIAL: NCT01321216
Title: ESTIMATION OF THE DISEASE BURDEN AND PREVALENT GENOTYPES OF ROTAVIRUS (RV) CAUSING GASTROENTERITIS (GE) IN CHILDREN <5 YEARS OF AGE IN LEBANON BASED ON A SENTINEL HOSPITAL-BASED SURVEILLANCE PROGRAM.
Brief Title: Rotavirus Burden and Genotypes in a Sentinel Hospital Surveillance System in Lebanon
Status: Completed | Type: Observational
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Makassed General Hospital (Other); Rafic Hariri University Hospital (Other); Hotel Dieu de France Hospital (Other); Hammoud Hospital University Medical Center (Other Government); Hopital Nini (Other); Nabatieh Governmental Hospital (Other)
Responsible Party: Principal Investigator, Dr. Ghassan Dbaibo, Pediatrician Doctor, American University of Beirut Medical Center
Other Study IDs: PED.GD.06
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-02

CONDITIONS: Gastroenteritis; Dehydration
Keywords: rotavirus; gastroenteritis; children; Pediatric; dehydration; vaccine
MeSH Terms: conditions — Gastroenteritis; Dehydration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples with rotavirus RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hospitalized Gastroenteritis: Children under 5 years of age hospitalized with gastroenteritis

SUMMARY:
This study aims to determine the contribution of rotavirus infection as a cause of gastroenteritis requiring hospitalization in children younger than 5 years of age. Additionally, a secondary aim will be to determine the genotypes of rotavirus that cause these infections as prevalent in Lebanon.

DETAILED DESCRIPTION:
This study will be performed at six large hospitals in Lebanon in the three largest cities Beirut, Tripoli, and Saida. The study will enroll children younger than 5 years of age who are admitted to the hospital because of gastroenteritis. Enrollment will continue for a period of two years at each hospital. Inclusion criteria are age < 5 years, with gastroenteritis as the main reason for admission to the hospital or for a stay in the Emergency Department longer than 12 hours. Exclusion criteria include onset of symptoms beyond 12 hours of admission (health-care associated infection). For all enrolled subjects, data will be collected about severity of illness, outcome, and history of vaccination. Stool samples will be collected for genotyping of rotavirus.

ELIGIBILITY:
Inclusion Criteria:

* Age < 5 years
* Gastroenteritis as admitting diagnosis
* Informed consent
* Parents willing and able to cooperate

Exclusion Criteria:

* Age > 5 years
* Onset of gastroenteritis beyond 12 hours of admission

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under 5 years of age admitted because of gastroenteritis to 6 major hospitals in Lebanon
Sampling Method: Non-Probability Sample
Enrollment: 1555 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Lebanon (4):
  - American University of Beirut, Beirut
  - Makassed General Hospital, Beirut
  - Rafik Hariri University Hospital, Beirut
  - Nini Hospital, Tripoli

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hospitalized Gastroenteritis
Started | 1555
Completed | 1555
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Children hospitalized with gastroenteritis
Arm/Group | Hospitalized Gastroenteritis
Number analyzed (Participants) | 1555
Age, Continuous [Mean (Full Range); unit: Months] | 22 [1 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 769
  Male | 786
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Lebanon | 1555

OUTCOME MEASURES:

1. Primary Outcome: Estimating the Incidence of Rotavirus Gastroenteritis Associated Hospitalization in Children < 5 Years of Age
Description: Incidence of rotavirus gastroenteritis associated hospitalization in children < 5 years of age was 30.3% by PCR
Time Frame: 2 years
Population: Children under 5 years of age hospitalized with gastroenteritis had a 30.3% rate of rotavirus infection
Measure: Count of Participants; unit: Participants
Arm/Group | Hospitalized Gastroenteritis
Number analyzed (Participants) | 1414
Participants | 428

2. Secondary Outcome: Identifying the Most Prevalent RV Genotypes in the Target Population Included in the Surveillance Program
Time Frame: 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Estimating the Proportion of Diarrheal Hospitalization Due to RV in Children < 5 Years of Age.
Time Frame: 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Determining the Age and Seasonal Distribution of RV Associated Hospitalizations in Children < 5 Years of Age
Time Frame: 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Determining Seasonal Changes and Year-to-year Changes With Respect to Predominant RV Genotypes
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Hospitalized Gastroenteritis
All-Cause Mortality (participants affected / at risk) | 0/1414
Serious Adverse Events (participants affected / at risk) | 0/1414
Other Adverse Events (participants affected / at risk) | 0/1414

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No